CLINICAL TRIAL: NCT00513643
Title: Pharmacodynamic and Pharmacokinetic Properties of Insulin Aspart: Dose - Ranging vs. Human Soluble Insulin
Brief Title: Metabolic Effect of Insulin Aspart and Human Insulin in Different Doses
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Profil Institut für Stoffwechselforschung GmbH (Industry)
Collaborators: Novo Nordisk A/S (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ISPS_Dose-ranging
Record Dates: First submitted 2007-08-08; First posted 2007-08-09 (Estimated); Last update posted 2007-08-09 (Estimated); Status verified 2007-08

CONDITIONS: Diabetes Mellitus
Keywords: euglycaemic glucose clamp; duration of action; late metabolic activity; hypoglycaemia
MeSH Terms: conditions — Diabetes Mellitus; Hypoglycemia | interventions — Insulin Aspart; Insulin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1 (Experimental): 6 U insulin aspart
  Interventions: Drug: insulin aspart
- 2 (Experimental): 12 U insulin aspart
  Interventions: Drug: insulin aspart
- 3 (Experimental): 24 U insulin aspart
  Interventions: Drug: insulin aspart
- 4 (Active Comparator): 6 IU human regular insulin
  Interventions: Drug: human regular insulin
- 5 (Active Comparator): 12 IU human regular insulin
  Interventions: Drug: human regular insulin
- 6 (Active Comparator): 24 IU human regular insulin
  Interventions: Drug: human regular insulin

INTERVENTIONS:
Drug: insulin aspart — 6, 12, 24 U s.c.
  Other Names: Novorapid
  Arms: 1; 2; 3
Drug: human regular insulin — 6, 12 and 24 IU sc
  Other Names: Actrapid
  Arms: 4; 5; 6

SUMMARY:
The metabolic effect of three different doses of insulin aspart and human insulin are investigated with the euglycaemic glucose clamp technique.

DETAILED DESCRIPTION:
Double-blind, randomized, 6-period cross-over study in 16 healthy subjects. Each patient participates in 6 euglycemic glucose clamp experiments each.

The time interval between the study days is 2 to 28 days. At the clamp visits, subjects are connected to a Biostator (MTB Medizintechnik, Ulm, Germany) and receive an intravenous human insulin infusion (rate of 0.15 mU/kg/min) over the duration of each experiment to prevent a rise in endogenous insulin secretion. After a baseline period of 2 h the trial drug (6, 12, or 24 U of either Insulin Aspart or regular human insulin in random order) are administered s.c. with a syringe into the abdominal wall. Glucose infusion rates (GIR) necessary to keep blood glucose concentrations close to the clamp level of 90 mg/dl (5 mmol/l) are administered and recorded by the Biostator every minute for a period of 12 h post-dosing. Blood samples are drawn at regular intervals for the analysis of C-peptide and (depending on the trial drug administered) serum insulin or serum Insulin Aspart concentrations (measured with specific ELISAs).

ELIGIBILITY:
Inclusion criteria:

* Signed informed consent obtained before any trial-related activities
* Healthy subjects between 18 and 45 years inclusive
* Considered generally healthy upon completion of medical history and physical examination
* Body mass index (BMI) < 27 kg/m2
* HbA1c < 6,1 %
* Non-smoker for at least three months
* Females of childbearing potential using acceptable methods of contraception, including tubal ligation, an intrauterine device (IUD), the oral contraceptive pill or barrier methods.

Exclusion Criteria:

* Participation in any other clinical trial and receipt of any investigational drug within four weeks prior to this trial
* Previous participation in this trial
* Clinically significant abnormal haematology or biochemistry screening test
* Any disease requiring use of non topical prescription medicines
* Any serious systemic infectious disease that occurred in the four weeks prior to the first dose of test drug
* Any intercurrent illness that may affect blood glucose
* Current addiction to alcohol or substances of abuse as determined by the investigator
* Known or suspected allergy against insulin or any component of the composition of the trial drug
* Blood donation > 500 ml within the last nine weeks
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or co-operation
* If female, subject is pregnant or lactating

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2002-04; Study Completion 2002-06 (Actual)

PRIMARY OUTCOMES:
AUC GIR 360-720 min | at each dosing (6 times during the trial)

SECONDARY OUTCOMES:
PK endpoints such as C max/ins, t max/ins, AUC ins 0-120 min, AUC ins 360-720 min, AUC ins 0-720 min | at each dosing visit (6 times during the study)
PD endpoints like GIR max, t max/GIR, AUC GIR 0-120 min, AUC GIR 0-720 min, t >2/GIR, early and late t 50%/GIR | at each dosing visit (6 times during the study)

CONTACTS AND LOCATIONS:
Overall Officials: Tim Heise, MD, Principal Investigator — Profil Institut für Stoffwechselforschung GmbH
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany

REFERENCES:
- See also: Profil Institut für Stoffwechselforschung — http://www.profil-research.de